CLINICAL TRIAL: NCT05147610
Title: Estimation of the Precision of the Icare200 in the Measurement of Intraocular Pressure in Comparison to the Gold Standard : Goldmann Applanation Tonometer
Brief Title: Precision of the Icare200 for Measuring Intraocular Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP 2021 COUTU; 2021-A00556-35 (Other: ANSM)
Record Dates: First submitted 2021-11-29; First posted 2021-12-07 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Glaucoma Eye
Keywords: Air puff tonometer; Goldmann tonometer; Applanation tonometer; Rebound tonometer; Icare 200; Comparative study; Intraocular pression

STUDY DESIGN:
Intervention Model Description: all participants receive the same intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients requiring an IOP (intra-Ocular Pression) measurement (Experimental): group representing adults patients in ophthalmologic consultation requiring an IOP measurement
  Interventions: Diagnostic Test: Intraocular pression

INTERVENTIONS:
Diagnostic Test: Intraocular pression — First, measurement of the eye pressure by air-puff tonometry and estimation of the pachymetries with the TONOREF III.
  Secondly, measurement of the eye pressure by GAT. Thirdly, measurement of the eye pressure by Icare 200.

SUMMARY:
In adult patients, intraocular pression readings are often taken with an air puff tonometer or goldmann tonometer. The current gold standard for IOP measurement is the Goldmann Applanation Tonometry (GAT). In some patients, measurement of intraocular pressure taken by applanation or by air puff may prove to be impossible for various reasons (obesity, handicap, mental disorder, blindness for Air Puff Tonometry, Anxiety, etc).

There are also many other devices that can be used to measure IOP, including those using rebound tonometry like the Icare 200.

The rebound tonometer would systematize IOP screening because of its ease of use, provided its measurements are reliable. In this prospective study, investigators will be measuring participant's IOP with Goldmann Applanation Tonometry, Icare 200 Tonometer and Air Puff Tonometry to see if there is an agreement in IOP between the different devices. Investigators will also look if there is a concordance between central corneal thickness and IOP. Moreover, investigators will look if there is a IOP concordance between the 3 different devices for hight BMI people. Indeed, higher body mass index tend to have difficulties with proper positioning at the slit lamp that may lead to inaccurate GAT measurements. Additionally, stress level of the patients with different tonometry devices will be recorded using a visual analog scale.

DETAILED DESCRIPTION:
Goldmann applanation tonometry remains the gold standard for intraocular pressure measurement in 2021. It provides the most exact approximation of true intraocular pressure based on Imbert Fick's law. The statistical normal (Gaussian distribution) of IOP is 15.8 plus or minus 5.14mmHg (2 standard deviations). Thus, an IOP value is considered to be pathological if it is greater than 21mmHg. In practice, the measurement with the Goldmann tonometer is done in a seated position due to the need to be installed behind a slit lamp. An anesthetic drop such as oxybuprocaine or tetracaine is instilled onto the ocular surface followed by a fluorescein drop. GAT may be associated with discomfort due to the need for topical anaesthesia which causes a burning sensation during about 30 secondes. Moreover, the patient must be compliant and the need to be seated makes measurement very difficult for some patients: pediatric, dementia, hight BMI or elderly people.

Rebound tonometers determine intraocular pressure by bouncing a small plastic tipped metal probe against the cornea.

As IOP increases, impact time decreases and rebound increases. It is portable, does not require the use of eye drops and is particularly suitable for children and non-cooperative patients. The examination is painless and can be performed without contact anesthesia. Different versions of tonometer using this principle exist. With the Icare 200 six measurements are taken. The 2 extreme values are eliminated and the average of the 4 remaining values gives the IOP.

In healthy subjects, the Icare tonometer gives results comparable to those of the Goldmann tonometer (1) with differences of less than 3 mmHg in 80% of cases (2).

In the literature, the type of rebound tonometer differs from that used in our study. Most of the previous studies compare the Icare RT01i, the Icare PRO, the Icare ONE, the Icare HOME or even the Icare 100 which are much older versions.

The Icare 200, the most recent model dating from 2018, has benefited from technical improvements. Intraocular pressure can be taken in any position.

Only one article in the literature has studied the diagnostic performance of Icare200 to date. In this study, Icare200 was compared with the Perkins tonometer in 2 groups of people, one group of healthy subjects and one group of patients with congenital glaucoma.

To date, we have no studies investigating the diagnostic performance of the iCare200 compared to the Goldmann tonometer. It is the interest of this study to compare the relationship of the IOP measurements obtained by Icare 200, Air Puff Tonometer and Goldmann Applanation Tonometry.

For this we have chosen to carry out a prospective study. We have chosen to include consenting adult patients consulting in ophthalmology consultation at Clermont-Ferrand University Hospital. This results in a large panel of patients with different IOP in order to observe enough IOP variability.

IOP measurements appear to correlate with corneal pachymetry (3). So, we chose to organize 4 subgroups according to pachymetry estimated by TONOREF III (high pachymetry, i.e. corneal thickness greater than 560um; low pachymetry, i.e. corneal thickness less than 500um; normal pachymetry, i.e. corneal thickness between 500 and 560um and subnormal pachymetry, i.e. corneal thickness between 500 and 520um).

Patient anxiety during tonometry will be measured using a visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

* Adult man ou woman who consults in ophthalmology for a reason justifying an IOP measurement
* Able to give informed consent
* Being affiliated with a social security system

Exclusion Criteria:

* Participants who are unable to have IOP measured by Goldmann Tonometry
* Participants who are unable to have IOP measured by air puff Tonometry
* Age younger than 18 years
* Inability to sit
* Corneal ulcer
* Refractive surgery
* Corneal Astigmatism >3D
* Participants who wear contact lenses
* Pregnancy
* Unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
mean difference (mmHg) between the Icare200 rebound tonometer and the Goldmann applanation tonometer | Day 0
  To evaluate the concordance of Goldmann tonometer and Icare 200 tonometer

SECONDARY OUTCOMES:
Diagnostic Performance | Day 0
  To evaluate the ability of detect ocular hypertension (>21mmHg)
Correlation between central corneal thickness and IOP | Day 0
  To evaluate the central corneal thickness on IOP measurement by Goldmann tonometer, Icare 200 tonometer and air puff tonometer
Effect of BMI on IOP | Day 0
  To compare IOP measurement between Goldmann tonometer, Air puff tonometer and Icare 200 tonometer depending of BMI (<29,9 ; 30-34,9 ; 35-39,9 ; >40)
Patient comfort during tonometry | Day 0
  To evaluate the discomfort felt by the patient after measurement by Icare 200 with a verbal scale

CONTACTS AND LOCATIONS:
Overall Officials: Adrien Coutu, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France